CLINICAL TRIAL: NCT00642382
Title: Randomized, Double Blind,Saline-Controlled, Multi-Center, Prospective Study to Evaluate the Safety and Effectiveness of Carticept's Agilus Device for the Treatment of Ankle Osteoarthritis
Brief Title: Safety and Effectiveness of Agilus (Hyaluronic Acid) for Ankle Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For safety concerns
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMI-CP-Ankle-001
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: OSTEOARTHRITIS
Keywords: Osteoarthritis; Hyaluronic Acid
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Agilus (Hyaluronic Acid)
  Interventions: Device: Agilus
- Control (Placebo Comparator): Normal Saline
  Interventions: Device: Normal saline

INTERVENTIONS:
Device: Agilus — Hyaluronic acid (Agilus)given by an intra-articular injection into the ankle for a total of 3 injections for 3 consecutive weeks.
  Other Names: Hyaluronic Acid
  Arms: Active
Device: Normal saline — Normal Saline given by an intra-operative injection into the ankle for a total of 3 injections for 3 consecutive weeks.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether Agilus is safe and effective in the treatment of mild to moderate ankle osteoarthritis.

DETAILED DESCRIPTION:
The objective of this study is to compare the safety and effectiveness of Agilus to a saline injection (control) in the treatment of mild to moderate ankle osteoarthritis. This is a multi-center, randomized, double blind, saline controlled, prospective study with two (2) treatment groups. The active group will receive one injection of Agilus per week for three consecutive weeks for a total of three injections. The control group will receive one injection of normal saline per week for three consecutive weeks for a total of three injections. Follow up visits will occur at 4 weeks, 12 weeks and 26 weeks following the third injection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chronic, unilateral ankle pain(i.e., in only one ankle) for at least 6 months
* Diagnosis of ankle OA confirmed by radiographs (X-ray)and clinical exam
* Are normally active, without aid of mobility devices(such as crutch, walker or cane)

Exclusion Criteria:

* Have used oral steroids within 30 days (inhaled or topical steroids are acceptable)
* Have received intra-articular injections of hyaluronic acid in any joint in the last 9 months
* Have received steroid injections in any joint in last 3 months
* Have had previous surgery or arthroscopy on the affected ankle in the last 12 months

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Baumhauer, MD, Principal Investigator — University of Rochester
Locations (19):
- United States (19):
  - Orthopaedic Associates of Hartford, Farmington, Connecticut
  - Pinnacle Research, Royal Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Institute For Foot and Ankle Reconstruction At Mercy, Baltimore, Maryland
  - Greater Chesapeake Orthopaedic Association, Baltimore, Maryland
  - Brigham Foot and Ankle Center, Boston, Massachusetts
  - Orthopedic Associates of Grand Rapids, Grand Rapids, Michigan
  - Minnesota Sports Medicine, Eden Prairie, Minnesota
  - University of Missouri, Columbia, Missouri
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - UMDNJ, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - Orthocarolina, Charlotte, North Carolina
  - Orthopedic Foot and Ankle Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Bone and Joint Clinic Houston, Houston, Texas
  - University of Texas Health Science Center At Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were not randomized and did not receive any intervention
Period: Overall Study
Arm/Group | Active | Control
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero patients were analyzed for this study due to the study being closed 2 months after it started. Baseline data were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
  <=18 years |  |  | 0
  Between 18 and 65 years |  |  | 0
  >=65 years |  |  | 0
Age, Continuous
Sex: Female, Male
  Female |  |  | 0
  Male |  |  | 0
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Comparison Between the Agilus Injection and the Saline Control Injection Groups in the Proportion of Subjects Experiencing a Reduction in the Assessment of Pain Determined by the AOS Subscale for Pain.
Time Frame: At 4, 12 and 26 weeks post 3rd injection
Population: Zero patients were analyzed for this study due to the study being closed 2 months after it started. Data were not collected
Arm/Group | Active | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Secondary Effectiveness Parameters That Will be Evaluated Include the Following That Evaluate Pain, Function, Subject's Global Assessment, Quality of Life and an Individual Subject Responder Analysis.
Time Frame: At 4, 12 and 26 weeks post 3rd injection
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months (study was closed prior to any data being collected)
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other